CLINICAL TRIAL: NCT07123506
Title: Beta-blockers for Prevention of Supraventricular Arrhythmia Following PFO Closure
Acronym: BRAVE PFO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2025-0005
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Atrial Fibrillation; Atrial Flutter; Tachycardia, Supraventricular; Heart Septal Defects, Atrial
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter; Tachycardia, Supraventricular; Heart Septal Defects, Atrial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beta-blocker treatment group (Experimental): After PFO closure, the beta-blocker treatment group will receive an extended-release beta-blocker, either bisoprolol or nebivolol, at a dose of 1.25 mg QD for 30 days.
  Interventions: Drug: Beta-blocker treatment group
- Non-treatment group (Experimental): After PFO closure, the non-treatment group will not receive a beta-blocker.
  Interventions: Drug: Non-treatment group

INTERVENTIONS:
Drug: Beta-blocker treatment group — After PFO closure, the beta-blocker treatment group will receive an extended-release beta-blocker, either bisoprolol or nebivolol, at a dose of 1.25 mg QD for 30 days.
  Arms: Beta-blocker treatment group
Drug: Non-treatment group — After PFO closure, the non-treatment group will not receive a beta-blocker.
  Arms: Non-treatment group

SUMMARY:
"The primary objective of the study is to evaluate whether the incidence of symptomatic or asymptomatic atrial fibrillation, atrial flutter, and atrial tachycardia within 30 days after percutaneous closure of idiopathic patent foramen ovale is reduced in the beta-blocker treatment group compared to the non-treatment group.

The secondary objective is to assess the safety and performance of the Cocoon Patent Foramen Ovale Occluder and collect real-world data on patient outcomes.

Patients will be randomly assigned in a 1:1 ratio to either the beta-blocker treatment group or the non-treatment group. Randomization will be performed using a 1:1 allocation ratio with stratification based on (1) PFO device size and (2) sex, employing a block randomization method (mixed block sizes of 4 or 6). This process will be conducted independently through an interactive web response system.

The beta-blockers used in this study are extended-release beta-blockers, specifically bisoprolol or nebivolol. The choice between bisoprolol and nebivolol will be determined at the discretion of the investigators, with the initial dose set at the minimum dose for each drug (1.25 mg once daily). During the study period, adjustments to the beta-blocker dose, including maintenance or modification, will be made based on the investigators' clinical judgment, taking into account the patient's heart rate, blood pressure, and medication adherence. All reasons for dose adjustments will be documented in detail."

ELIGIBILITY:
Inclusion Criteria:

1. Age 19 years or older
2. Patients scheduled to undergo Patent Foramen Ovale closure using the Cocoon Patent Foramen Ovale Occluder
3. Individuals who have provided informed consent for study participation

Exclusion Criteria:

1. History of paroxysmal, persistent, or permanent atrial arrhythmia
2. Atrial arrhythmia confirmed by a 14-day Holter ECG using the AT Patch before PFO closure
3. Patients with uncontrolled asthma or chronic obstructive pulmonary disease (COPD)
4. Patients with high-degree atrioventricular (AV) block
5. History of heart failure, severe valvular disease, or left ventricular dysfunction (ejection fraction <50%)
6. Patients for whom initiating or discontinuing beta-blocker therapy is deemed impossible by the investigator
7. Patients who, as assessed by the investigator, cannot be followed up for one year after enrollment
8. Patients with hypersensitivity or contraindications to any proposed drug therapy or device component
9. Patients with an expected life expectancy of less than one year
10. Patients currently participating in another investigational drug or device study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2029-05-03 (Estimated)

PRIMARY OUTCOMES:
Atrial Arrhythmias Within 30 Days After PFO Closure | Within 30 days after Patent Foramen Ovale closure
  The occurrence of at least one episode of symptomatic or asymptomatic atrial fibrillation, atrial flutter, or atrial tachycardia lasting 30 seconds or longer within 30 days after PFO closure. Monitoring will be conducted using a 14-day Holter ECG with the AT Patch during the initial 14 days, followed by an additional clinical assessment and ECG evaluation on day 15.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Cardiovascular Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No